CLINICAL TRIAL: NCT03079388
Title: Randomized Control Trial of the Use of Supplementary Food and Measures to Control Inflammation in Malnourished Pregnant Women to Improve Birth Outcomes
Brief Title: Nutritional and Anti-infective Interventions for Malnutrition in Pregnancy (Beleuman Welbodi)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: The Children's Investment Fund Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 201611119
Record Dates: First submitted 2017-03-05; First posted 2017-03-14 (Actual); Last update posted 2021-01-07 (Actual); Status verified 2021-01

CONDITIONS: Pregnancy; Malnutrition in Pregnancy; Nutrition Disorders; Stunting
MeSH Terms: conditions — Nutrition Disorders; Growth Disorders | interventions — fanasil, pyrimethamine drug combination; Insecticide-Treated Bednets; Azithromycin; Albendazole; Therapeutics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ready-to-use supplementary food + anti-infective bundle (Experimental): The women randomized to this arm will receive a ready-to-use-supplementary food (RUSF) designed specifically for pregnancy. The RUSF will provide a total of 520 kcal, 18 g protein, and 200% of recommended daily allowance (RDA) for most micronutrients during pregnancy. The supplement is also optimized to provide excellent protein quality and optimal polyunsaturated fatty acid composition. These women will receive 5 anti-infective interventions: 1) insecticide-treated mosquito net, 2) monthly intermittent preventive treatment of malaria during pregnancy (IPTp) 3) azithromycin at the second and third trimester 4) albendazole given in second trimester, and 5) bacterial vaginosis testing and treatment at enrollment and again at weeks 28-34
  Interventions: Dietary Supplement: Ready-to-use-supplementary food; Drug: Monthly intermittent preventive treatment of malaria during pregnancy (IPTp); Other: Insecticide-treated mosquito net; Drug: Azithromycin; Drug: Albendazole; Combination Product: Bacterial vaginosis testing and treatment
- Corn-soy-blend (Active Comparator): The women randomized to this arm will receive the standard of care for Sierra Leone. The treatment provided to women in this group includes 3.5 kg super cereal with 350 g vegetable oil every two weeks. This provides 250 mg portion/day of the super cereal and 25g oil/day for the mother. Women will receive the food for the duration of their pregnancy. These women will receive the current recommendations of the government of Sierra Leone, which includes standard intermittent preventive treatment of malaria during pregnancy (IPTp) of 2 doses of sulfadoxine/ pyrimethamine, iron and folic acid supplement with a goal of 90 pills/pregnancy, an insecticide-treated mosquito net, and albendazole for deworming in the second trimester.
  Interventions: Dietary Supplement: Corn-soy-blend; Drug: Standard intermittent preventive treatment of malaria during pregnancy (IPTp); Other: Insecticide-treated mosquito net; Drug: Albendazole

INTERVENTIONS:
Dietary Supplement: Ready-to-use-supplementary food — Specially formulated supplementary food for pregnancy
  Arms: Ready-to-use supplementary food + anti-infective bundle
Dietary Supplement: Corn-soy-blend — Standard of care for malnutrition in pregnancy in Sierra Leone
  Arms: Corn-soy-blend
Drug: Monthly intermittent preventive treatment of malaria during pregnancy (IPTp) — Sulfadoxine-pyrimethamine (500 mg / 25 mg) given every 4 weeks, beginning at enrollment or at 13 weeks' gestation, whichever is later.
  Other Names: Sulfadoxine-pyrimethamine
  Arms: Ready-to-use supplementary food + anti-infective bundle
Drug: Standard intermittent preventive treatment of malaria during pregnancy (IPTp) — Standard of care for Sierra Leone is 2 doses of sulfadoxine/ pyrimethamine (500mg/ 25mg).
  Other Names: Sulfadoxine-pyrimethamine
  Arms: Corn-soy-blend
Other: Insecticide-treated mosquito net — An insecticide-treated mosquito net at the time of enrollment into the study.
Drug: Azithromycin — Azithromycin 1 gram given once in second trimester and again during weeks 28-34 of gestation.
  Arms: Ready-to-use supplementary food + anti-infective bundle
Drug: Albendazole — Single dose albendazole 400mg given in the second trimester.
Combination Product: Bacterial vaginosis testing and treatment — Testing for bacterial vaginosis at enrollment and again at weeks 28-34 using a rapid diagnostic test for sialidase. Those with positive tests will receive extended release metronidazole 750mg daily for 7 days.
  Arms: Ready-to-use supplementary food + anti-infective bundle

SUMMARY:
Acute malnutrition in pregnancy is a risk factor for adverse outcomes in mothers and their unborn children. Undernutrition during pregnancy can result in maternal complications such as life-threatening hemorrhage and hypertensive disorders of pregnancy and infant complications such as intrauterine growth retardation, low birth weight, pre-term delivery and poor cognitive development. Poor women in the developing world are at heightened risk of malnutrition due to inadequate dietary intake and are subject to transmission of a number of infections including malaria, intestinal helminths, and genitourinary infections. Food interventions for malnutrition may be less effective under conditions with excessive inflammation and infection, and especially so during pregnancy. Without specifically addressing treatment for infections, undernourished mothers may be less responsive to nutritional interventions. The benefits of treating both malnutrition and common infections simultaneously remain largely unstudied. This study tests the hypothesis that malnourished pregnant women receiving 100 grams per day of a specially formulated ready-to-use supplementary food in addition to a combination of 5 anti-infective interventions will have greater weight gain in pregnancy and deliver larger, longer infants than women receiving the standard of care. The outcome of the pregnancy and maternal nutritional status will be followed until 6 months after delivery.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women and consenting to study participation
* Fundal height not greater than 32 cm
* Mid-upper arm circumference ≤23 cm
* Planning to reside in the study area during pregnancy and 6 months post partum
* Attending 1 of the 40 antenatal clinic sites

Exclusion Criteria:

* < 16 years of age without adult willing to consent
* Known pregnancy complications such as gestational diabetes, pre-eclampsia, hypertension

Min Age: 14 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Must be pregnant woman
Enrollment: 1489 (Actual)
Dates: Start 2017-02-27 (Actual); Primary Completion 2019-09-24 (Actual); Study Completion 2020-02-24 (Actual)

PRIMARY OUTCOMES:
Infant birth length | up to 40 weeks
  mean birth length of infants born to mothers in the study

SECONDARY OUTCOMES:
Maternal weight gain | up to 40 weeks
  Average weekly weight gain of women in the study
Proportion recovered from maternal malnutrition | up to 40 weeks
  proportion of women who reach mid-upper-arm circumference (MUAC) > 23 cm
Premature delivery | up to 36 weeks
  proportion of infants born prematurely
Newborn head circumference | up to 40 weeks
  mean head circumference of infants born to women in the study
Infant birth weight | up to 40 weeks
  mean birth weights of infants born to mothers in the study
Infant weight at 6 weeks, 3 and 6 months | up to 6 months
  infant ponderal growth
Infant length at 6 weeks, 3 and 6 months | up to 6 months
  infant linear growth
Infant survival at 3 and 6 months | up to 6 months
  survival of infants in the study

CONTACTS AND LOCATIONS:
Overall Officials: Mark J Manary, MD, Study Chair — Washington University School of Medicine
Locations (1):
- 1 Moriba Street, Pujehun, Pujehun District, Sierra Leone

REFERENCES:
- [Derived] Hendrixson DT, Lasowski PN, Koroma AS, Manary MJ. Newborn Mid-Upper Arm Circumference Identifies Low-Birth Weight and Vulnerable Infants: A Secondary Analysis. Curr Dev Nutr. 2022 Sep 12;6(10):nzac138. doi: 10.1093/cdn/nzac138. eCollection 2022 Oct. PMID 36475019
- [Derived] Hendrixson DT, Smith K, Lasowski P, Callaghan-Gillespie M, Weber J, Papathakis P, Iversen PO, Koroma AS, Manary MJ. A novel intervention combining supplementary food and infection control measures to improve birth outcomes in undernourished pregnant women in Sierra Leone: A randomized, controlled clinical effectiveness trial. PLoS Med. 2021 Sep 28;18(9):e1003618. doi: 10.1371/journal.pmed.1003618. eCollection 2021 Sep. PMID 34582451
- [Derived] Hendrixson DT, Koroma AS, Callaghan-Gillespie M, Weber J, Papathakis P, Manary MJ. Use of a novel supplementary food and measures to control inflammation in malnourished pregnant women in Sierra Leone to improve birth outcomes: study protocol for a prospective, randomized, controlled clinical effectiveness trial. BMC Nutr. 2018 Apr 2;4:15. doi: 10.1186/s40795-018-0218-y. eCollection 2018. PMID 32153879